CLINICAL TRIAL: NCT05646290
Title: Validation of a Machine Learning Model for Predicting Anastomotic Leakage of Esophagogastrostomy and Esophagojejunostomy: A Multicenter Prospective Study
Brief Title: Validation of a Model for Predicting Anastomotic Leakage
Status: Completed | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20211255
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: machine learning; anastomotic leakage; total and proximal gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will validate a machine learning model for predicting anastomotic leakage of esophagogastrostomy and esophagojejunostomy.

DETAILED DESCRIPTION:
Anastomotic leakage is a fatal complication after total and proximal gastrectomy in gastric cancer patients. Identifying patients with high-risk of AL is important for guiding the surgeons' decision making, such as a more rigorous anastomotic operation， placing a jejunal feeding tube and dual-lumen flushable drainage catheter. We have developed a high-performance machine learning model based on 1660 gastric cancer patients, which showed good discrimination of anastomotic leakage. Hence, this multi-center prospective study will validiate the usability of the model for predicting anastomotic leakage in gastric cancer patients who receive total and proximal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years.
2. Primary gastric adenocarcinoma confirmed by preoperative pathology.
3. Expected curative resection via total or proximal gastrectomy.
4. American Society of Anesthesiologists (ASA) class I, II, or III.
5. Written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Severe mental disorder or language communication disorder.
3. Other surgical procedures of gastrectomy is performed.
4. Interrupted of surgery for more than 30 minutes due to any cause.
5. Malignant tumors with other organs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients undergoing total or proximal gastrectomy in five medical centers (Tongji Hospital, Wuhan No. 1 Hospital, Xianning Central Hospital, Huanggang Central Hospital and Jingzhou Central Hospital) are included in this perspective study.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of anastomotic leakage | Within 30 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China